CLINICAL TRIAL: NCT06880055
Title: Shield Post-Approval Study Protocol
Acronym: SOLAR
Status: Recruiting | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-GI-003
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Colo-rectal Cancer
Keywords: Screening; Shield
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Enrolled Subjects: Subjects age 45 to 81 at average risk of CRC who meet inclusion, do not meet exclusion criteria, and who successfully enroll in the study.
  Interventions: Diagnostic Test: Shield Blood Test for colo-rectal cancer Screening

INTERVENTIONS:
Diagnostic Test: Shield Blood Test for colo-rectal cancer Screening — Shield Blood Test for colo-rectal cancer Screening

SUMMARY:
The Shield post-approval study (PAS) is a prospective, longitudinal study supplemented with Real World Evidence (RWE) to evaluate the longitudinal performance of Shield in an average risk population at a second round of testing for individuals between the ages of 45 and 81 at average risk of CRC using colonoscopy as the reference method.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the fourth most diagnosed cancer and second leading cause of cancer-related death in the US, with an estimated 53,010 deaths attributable to CRC in 2024. The risk of CRC increases with age, with the majority of cases and deaths occurring in individuals aged 65 years or older. While the incidence of CRC in Americans 65 years of age or older has decreased over the last decade, the incidence of CRC in younger Americans aged 55 years or younger has been increasing since the mid-1990s. CRC disproportionately affects minority populations, with American Indian/Alaska Native and Black/African American populations having the highest incidence and mortality rates1; this is further exacerbated by systemic barriers to current CRC screening options.

CRC primarily arises from a precursor lesion, the adenomatous polyp (i.e., adenoma), that grows from the epithelial cells of the colorectal mucosa. Adenomas that grow larger than 10 mm or have elements indicating a risk of malignant transformation (e.g., high-grade dysplasia or villous features) are defined as advanced adenomas (AAs). The vast number of adenomas, even those with features classifying them as AAs, do not progress into a colorectal malignancy. Colonoscopy cannot always distinguish adenomas or advanced adenomas from other polyp histology; thus, polypectomy is routinely performed for lesions identified on endoscopy. The transition rate from adenoma onset to CRC development is estimated to be 12.5 to 25 years. This slow transition from adenoma onset to CRC onset allows for multiple CRC screening opportunities over a lifetime, providing the ability to intervene along the disease development course and the potential to detect and remove adenomas, prevent colorectal cancer, and reduce CRC incidence and subsequently, disease mortality.

Once CRC has developed, tumor staging is consistent with other solid tumors and defined based on how far the cancer has spread within the body. In Stage 0 (carcinoma in situ), the cancer cells are only in the colorectal mucosa. In Stage I, the cancer has spread to the muscular layer of the colorectum but not to nearby tissue or lymph nodes. In Stage II, the cancer has grown through the wall of the colorectum and potentially to nearby tissues but has not spread to nearby lymph nodes. In Stage III, the cancer has spread to nearby lymph nodes but not to distant parts of the body. In Stage IV, the cancer has spread to one or more distant parts of the body. The estimated time frame from CRC onset to a symptomatic diagnosis of CRC is estimated to be 4-5 years, in the absence of early detection through asymptomatic cancer screening. Tumor size and location can influence the rate of transition through the stages of CRC. The 5-year survival rate for localized disease (Stage I-II) is 91%, and is 72% for regional disease (Stage III), while the 5-year survival for metastatic disease (Stage IV) is only 14%. These statistics highlight the ability to reduce CRC-related mortality by detection of early-stage (Stage I-III) disease where therapeutic intervention has the potential to result in a cure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 45-81 years at time of consent
2. Intending to undergo a standard of care Shield test
3. Considered by a physician or healthcare provider as being of 'average risk' for CRC; 'Average-risk' individuals in the context of CRC screening are defined as those who do not have symptoms of CRC and do not have increased risk factors for the disease (i.e., prior diagnosis of CRC, adenomatous polyps, or inflammatory bowel disease; family history of CRC or known hereditary predisposition to CRC).
4. Subject agrees to comply with study procedures and associated standard of care assessments.

Exclusion Criteria:

1. Undergoing colonoscopy for investigation of symptoms
2. Personal history of colorectal cancer (CRC), adenomas, or other related cancers
3. Family history of CRC, defined as having one or more first-degree relative (parent, sibling, or child) diagnosed with CRC at any age
4. Positive result on another colorectal cancer screening method within the last six months, or:

   * 12 months for fecal occult blood test (FOBT) or fecal immunochemical test (FIT)
   * 36 months for FIT-DNA test
5. Personal history of any of the following high-risk conditions for colorectal cancer:

   * Inflammatory Bowel Disease (IBD), including chronic ulcerative colitis (CUC) and Crohn's disease
   * Familial adenomatous polyposis (FAP)
   * Other hereditary cancer syndromes including but not limited to:

     * Hereditary non-polyposis colorectal cancer syndrome (HNPCC) or "Lynch Syndrome", Peutz- Jeghers Syndrome, MUTYH Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis
6. Positive Shield test result within the previous 3 years
7. History of any malignancy (patients who have undergone surgical removal of skin squamous cell cancer may be enrolled provided the procedure was completed at least 12 months prior to the date of provision of informed consent for the study)
8. Known diagnosis of inflammatory bowel disease
9. Currently taking any anti-neoplastic or disease-modifying anti-rheumatic drugs (DMARDs)
10. Any major physical trauma (e.g., disruption of tissue, surgery, organ transplant, blood product transfusion) within the 30 days leading up to the provision of informed consent
11. Known medical condition which, in the opinion of the Investigator, should preclude enrollment into the study
12. Participation in a clinical research study in which an experimental medication has been administered or may be administered within the 30 days leading up to providing informed consent or may be administered through the time of colonoscopy

Ages: 45 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects age 45 to 81 at average risk of CRC who meet inclusion, do not meet exclusion criteria, and who successfully enroll in the study
Sampling Method: Probability Sample
Enrollment: 3375 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Performance measures of the Shield test will be assessed for the second testing interval | 33-42 Months Post-Enrollment
  * Advanced Neoplasia Specificity
  * AA Sensitivity
  * CRC Sensitivity
  * PPV for: CRC, AA, and advanced neoplasia.
  * NPV for: CRC and advanced neoplasia

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Southeast Valley Gastroenterology Consultants, Chandler, Arizona
  - Southeast Valley Gastroenterology Consultants, Gilbert, Arizona
  - Alliance Research Institute, LLC, Canoga Park, California
  - Paragon Rx Clinical, Inc., Garden Grove, California
  - Amicis Research Center, Granada Hills, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Digestive Disease Associates, Branford, Connecticut
  - Gastroenterology Consultants of Boca Raton, LLC, Boca Raton, Florida
  - Physicians Group of South Florida, North Miami, Florida
  - Digestive Disease Consultants, Bourbonnais, Illinois
  - Christie Clinic, Champaign, Illinois
  - GI Solutions of Illinois, Chicago, Illinois
  - Digestive Health Services, Downers Grove, Illinois
  - Gastroenterology and Internal Medicine Specialists (GAIMS), Lake Barrington, Illinois
  - Southwest Gastroenterology (SWG), Oak Lawn, Illinois
  - Hutchinson Clinic, Hutchinson, Kansas
  - Northlake Gastroenterology Associates, Covington, Louisiana
  - Northlake Gastroenterology Associates, Hammond, Louisiana
  - Gastroenterology Associates of New Jersey, LLC, Clifton, New Jersey
  - Gastroenterology Associates of New Jersey, Hackensack, New Jersey
  - Gastroenterology Associates of New Jersey, LLC, Montclair, New Jersey
  - Gastroenterology Associates of New Jersey, LLC, Ridgewood, New Jersey
  - Gastroenterology Associates of New Jersey, LLC, Wayne, New Jersey
  - Gastroenterology Associates of New Jersey, Wayne, New Jersey
  - Associated Gastroenterologists of Central New York, Camillus, New York
  - Syracuse Gastroenterological Associates, P.C., East Syracuse, New York
  - Associated Gastroenterologists of Central New York, Fayetteville, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - GastroCare LI, Valley Stream, New York
  - Cary Gastroenterology Associates, Cary, North Carolina
  - Piedmont Healthcare, P.A., Mocksville, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Sanford Cardiology Pinehurst Medical Clinic, Sanford, North Carolina
  - Piedmont Healthcare LLC, Statesville, North Carolina
  - US Digestive Health at Blair, Altoona, Pennsylvania
  - Health Living at Pottstown Medical Specialists, Inc, Pottstown, Pennsylvania
  - Premier Family Physicians, Austin, Texas
  - Integrity Advanced Therapeutics, PLLC, Houston, Texas
  - Center for Digestive Disease, Shenandoah, Texas
  - Horizon Clinical Research Group, Tomball, Texas
  - Tidewater Physician Multispecialty Group Clinical Research, Williamsburg, Virginia

IPD SHARING:
Plan to Share IPD: No